CLINICAL TRIAL: NCT02527681
Title: An Open-label Study to Evaluate the Single-dose Pharmacokinetics and Safety of Ceftobiprole in Neonate and Infant Subjects Aged up to 3 Months Undergoing Treatment With Systemic Antibiotics
Brief Title: Pharmacokinetics and Safety of Ceftobiprole in Neonates and Infants up to 3 Months Treated With Systemic Antibiotics
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: on July 07, 2020 due to slow enrollment; there were no safety concerns.
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPR-PIP-001; 2013-004614-18 (EudraCT Number)
Record Dates: First submitted 2015-08-05; First posted 2015-08-19 (Estimated); Results first posted 2021-01-06 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — ceftobiprole medocaril; ceftobiprole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ceftobiprole (Experimental): Ceftobiprole medocaril is the water-soluble prodrug of ceftobiprole, an advanced-generation cephalosporin developed for intravenous administration. Ceftobiprole is characterized by potent, broad-spectrum antimicrobial activity against both Gram-positive and Gram-negative pathogens.
  Interventions: Drug: Ceftobiprole medocaril

INTERVENTIONS:
Drug: Ceftobiprole medocaril — Ceftobiprole medocaril was administered as a single intravenous infusion, with a bodyweight-adjusted volume, at a constant rate over 4 hours. The ceftobiprole dose was 7.5 mg/kg, which corresponds to 10.0 mg ceftobiprole medocaril.
  Other Names: ceftobiprole

SUMMARY:
This study characterized the pharmacokinetics and safety of a single dose of ceftobiprole in neonates and infants aged ≤ 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Neonates and infants ≤3 months, with gestational age ≥28 weeks
* Documented or presumed (or at risk of) bacterial infections, and currently receiving antibiotic treatment
* Expected to survive beyond the first 7 days after enrollment
* Sufficient vascular access to receive study drug, and to allow blood sampling at a site separate from the study drug infusion site
* Parent's / legally acceptable representative's informed consent to participate in the study

Exclusion Criteria:

* Major birth defect or malformation syndrome
* Proven presence of an immunodeficiency
* HIV or other congenital viral or fungal infection
* Significant laboratory abnormalities including: hematocrit <20%; absolute neutrophil count <0.5x10⁹/L; platelet count < 50x10⁹/L; alanine aminotransferase or aspartate aminotransferase >3 times the age-specific upper limit of normal
* Impaired renal function or known significant renal disease
* Any condition which would make the subject or caregiver, in the opinion of the investigator, unsuitable for the study

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Engelhardt, MD, Study Director — Basilea Pharmaceutica
Locations (14):
- United States (9):
  - Loma Linda University Medical Center, Loma Linda, California
  - University of Southern California, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Beacon Children's Hospital, South Bend, Indiana
  - Norton Children's Hospital, Louisville, Kentucky
  - Duke University Hospital, Durham, North Carolina
  - University of Pittsburgh Medical Center Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - West Virginia University School of Medicine, Morgantown, West Virginia
- UZ Leuven, Leuven, Belgium
- Klinikum der Universität München, Munich, Germany
- Children Clinical University Hospital, Riga, Latvia
- Vilnius University Children's Hospital, Vilnius, Lithuania
- University Children's Hospital of Kraków, Krakow, Poland

REFERENCES:
- [Derived] Rubino CM, Polak M, Schropf S, Munch HG, Smits A, Cossey V, Tomasik T, Kwinta P, Snariene R, Liubsys A, Gardovska D, Hornik CD, Bosheva M, Ruehle C, Litherland K, Hamed K. Pharmacokinetics and Safety of Ceftobiprole in Pediatric Patients. Pediatr Infect Dis J. 2021 Nov 1;40(11):997-1003. doi: 10.1097/INF.0000000000003296. PMID 34533489

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects with documented or presumed bacterial infection receiving standard-of-care antibiotic treatment were screened.
Groups:
- Ceftobiprole ITT/Safety Population: All subjects who received any quantity of study drug.
Period: Overall Study
Arm/Group | Ceftobiprole ITT/Safety Population
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ceftobiprole ITT/Safety Population
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 13 [8 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: The maximum observed plasma concentration (Cmax)
Time Frame: Blood samples for pharmacokinetic (PK) analysis were obtained pre-dose, and at 2, 4, 6, 8, and 12 hours after the start of dosing.
Measure: Median (Full Range); unit: μg/mL
Groups:
- Ceftobiprole PK Population: All subjects who received study drug and had adequate samples for determination of time-plasma concentration profiles of ceftobiprole.
Arm/Group | Ceftobiprole PK Population
Number analyzed (Participants) | 13
μg/mL | 11.2 [8.68 to 32.6]

2. Primary Outcome: Tmax
Description: The time of maximum observed plasma concentration (Tmax)
Time Frame: Blood samples for PK analysis were obtained pre-dose, and at 2, 4, 6, 8, and 12 hours after the start of dosing.
Measure: Median (Full Range); unit: hours
Arm/Group | Ceftobiprole PK Population
Number analyzed (Participants) | 13
hours | 4.00 [4.00 to 4.00]

3. Primary Outcome: AUC0-last
Description: The area under the plasma concentration-time curve from time zero to the time of the last measurable concentration (AUC0-last)
Time Frame: Blood samples for PK analysis were obtained pre-dose, and at 2, 4, 6, 8, and 12 hours after the start of dosing.
Measure: Median (Full Range); unit: μg•hours/mL
Arm/Group | Ceftobiprole PK Population
Number analyzed (Participants) | 13
μg•hours/mL | 60.6 [49.1 to 126.0]

4. Primary Outcome: T>MIC of 4 mg/L
Description: The duration of time after dose for which free-drug concentrations remained above a value of 4 mg/L (T>MIC of 4 mg/L)
Time Frame: Blood samples for PK analysis were obtained pre-dose, and at 2, 4, 6, 8, and 12 hours after the start of dosing.
Measure: Median (Full Range); unit: hours
Arm/Group | Ceftobiprole PK Population
Number analyzed (Participants) | 13
hours | 5.40 [3.77 to 8.13]

ADVERSE EVENTS:
Time Frame: After start of study drug administration through the follow-up visit at study Day 7±3, relevant worsening of a subject's status was to be recorded as an adverse event (AE).
Description: Once an AE was detected, it was proactively followed up at each visit (or more frequently if necessary) for any changes in severity, relationship to the study drug, interventions required for treatment, and the event's outcome. Serious adverse events (SAEs) were to be additionally reported and recorded on SAE report forms.
Arm/Group | Ceftobiprole ITT/Safety Population
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 4/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftobiprole ITT/Safety Population (N=15)
Diaphragmatic hernia (Gastrointestinal disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftobiprole ITT/Safety Population (N=15)
Drug Dependence (Psychiatric disorders) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT02527681/Prot_001.pdf
  • Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT02527681/SAP_000.pdf